CLINICAL TRIAL: NCT05150795
Title: The Effect of Preoperative Oral Pregabalin and Intraoperative Fentanyl on Postoperative Analgesia in Diagnostic Laparoscopic Gynecologic Surgery: a Comparative Study
Brief Title: Effect of Preoperative Oral Pregabalin Versus Intraoperative Fentanyl on Postoperative Analgesia
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ghada M.Samir, Assistant Professor of Anesthesia, Intensive care and Pain Management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R18/2020/2021
Record Dates: First submitted 2021-10-08; First posted 2021-12-09 (Actual); Last update posted 2025-01-29 (Actual); Status verified 2025-01

CONDITIONS: Post Operative Pain, Acute
Keywords: pregabalin; analgesia
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group Pregabalin (Active Comparator): Patients will receive oral pregabalin capsule (150 mg) 90 min before induction of anesthesia, and will receive a bolus injection of 10 ml saline at induction of anesthesia
  Interventions: Drug: Pregabalin 150mg
- Group Fentanyl (Active Comparator): Patients will receive oral placebo capsule identical to the trial drug in size, shape and color, 90 min before induction of anesthesia and will receive a bolus injection of 10 ml of 1µg /kg fentanyl at induction of anesthesia
  Interventions: Drug: Fentanyl 100 micrograms ampoule

INTERVENTIONS:
Drug: Pregabalin 150mg — Compare the postoperative analgesic effect of pre-operative oral pregabalin (Study group), to the intraoperative intravenous fentanyl (Control group) in diagnostic laparoscopic gynecologic surgery.
  Arms: Group Pregabalin
Drug: Fentanyl 100 micrograms ampoule — Compare the postoperative analgesic effect of pre-operative oral pregabalin (Study group), to the intraoperative intravenous fentanyl (Control group) in diagnostic laparoscopic gynecologic surgery.
  Arms: Group Fentanyl

SUMMARY:
Pregabalin is a structural analogue of gamma amino butyric acid (GABA). It binds to presynaptic alpha-2-delta subunit of voltage gated calcium channels in the brain and the spinal cord. Thus, it modulates the release of excitatory neurotransmitters, such as glutamate, norepinephrine, substance-P, and calcitonin gene related peptide. Also, it causes inhibitory modulation of overexcited neurons and restores them to a normal state.

Pre-emptive analgesia aims to reduce postoperative opioid consumption especially in ambulatory surgeries. Pregabalin (PGB) is an emerging drug in this field. Different doses of preoperative oral pregabalin (75, 150 and 300 mg) are described in the literature with a dose-response analgesic relationship and reduction of opioid use; however increasing the dose results in increasing the incidence of side effects mainly sedation and dizziness.

Perioperative use of opioids for analgesia may result in side effects; like nausea, vomiting, excessive sedation, respiratory depression, pruritus, and urinary retention.The concomitant use of opioids with pregabalin may result in excess sedation and somnolence, so, the use of opioids with pregabalin should be limited to patients with inadequate alternative options.

DETAILED DESCRIPTION:
Our study aims to compare the postoperative analgesic effect of pre-operative oral pregabalin (Study group), to the intraoperative intravenous fentanyl (Control group) in diagnostic laparoscopic gynecologic surgery.

Patienrs will be selected by simple randomization by computer generated system. Pregabalin 150 mg oral capsule and a placebo capsule will be available on the morning of operation.

Also, 2 syringes of 10 ml volumes will be prepared; the first contains normal saline and the second contains the fentanyl dose of 1 µg /kg calculated according to the patient's body weight and diluted to a 10 ml volume.

Patients will then be divided into 2 equal groups of 40 patients each:

Group P: Patients will receive oral pregabalin capsule (150 mg) 90 min before induction of anesthesia, and will receive a bolus injection of 10 ml saline at induction of anesthesia.

Group F: Patients will receive oral placebo capsule identical to the trial drug in size, shape and color, 90 min before induction of anesthesia and will receive a bolus injection of 10 ml of 1µg /kg fentanyl at induction of anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I

Exclusion Criteria:

* Patients' refusal
* use of sedatives, hypnotics, anti-psychotic or antidepressant drugs
* history of drug/alcohol abuse
* history of chronic pain
* daily intake of analgesics
* history of epilepsy

Ages: 21 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 80 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Changes in post-operative pain score at rest over time | 1 hour
  Intensity of pain will be monitored at 15 and 30min after arrival to the PACU, then 1h before discharge from the PACU. For analysis, pain severity will be categorized as absent (VAS=0), mild (VAS=1-3), moderate (VAS=4-7), severe (VAS=7-9), and very severe (VAS=10).
Changes in post-operative pain score on coughing over time | 1 hour
  Intensity of pain will be monitored at 15 and 30min after arrival to the PACU, then 1h before discharge from the PACU. For analysis, pain severity will be categorized as absent (VAS=0), mild (VAS=1-3), moderate (VAS=4-7), severe (VAS=7-9), and very severe (VAS=10).

SECONDARY OUTCOMES:
Pre-operative level of patient sedation assessed by the sedation score | 1 hour
  assessed 1 hour after administering the oral capsules by the sedation score from 0 to 4. 0=Awake and agitated, 1= Awake and comfortable, 2= Asleep and arousable, 3= Asleep with sluggish response to verbal commands or touch, 4= No response to verbal command or touch.
Duration of surgery | 2 hours
  Measured in minutes
Duration of anesthesia | 3 hours
  Measured in minutes
mean values of systolic blood pressure (SBP) | 4 hours
  mean values of SBP at pre-operative baseline, before induction of anesthesia, 5min after endotracheal intubation, before pneumoperitoneum, during the first 30 minutes (at 10, 20 and 30 min) of pneumoperitoneum, after release of pneumoperitoneum and 10 min after extubation in the PACU
Intra-operative additional doses of fentanyl given | 3 hours
  Rescue analgesia needed in micrograms
Postoperative level of patient sedation | 1 hour
  assessed by the sedation score from 0 to 4. 0=Awake and agitated, 1= Awake and comfortable, 2= Asleep and arousable, 3= Asleep with sluggish response to verbal commands or touch, 4= No response to verbal command or touch.
Post-operative pain score | 12 hours
  at rest and on coughing using the Visual Analogue Score (VAS) score from 0 to 10 where 0= no pain and 10 is the worst pain felt. Pain severity will be categorized as absent (VAS=0), mild (VAS=1-3), moderate (VAS=4-7), severe (VAS=7-9), and very severe (VAS=10).
Pethidine requirements | 1 hour
  Number of patients requiring pethidine in the PACU
sPO2 | 4 hours
  recorded in the induction room and in the PACU
changes in mean values of diastolic blood pressure (DBP) | 4 hours
  mean values of DBP at pre-operative baseline, before induction of anesthesia, 5min after endotracheal intubation, before pneumoperitoneum, during the first 30 minutes (at 10, 20 and 30 min) of pneumoperitoneum, after release of pneumoperitoneum and 10 min after extubation in the PACU
changes in mean values of mean blood pressure (MBP) | 4 hours
  mean values of MBP,at pre-operative baseline, before induction of anesthesia, 5min after endotracheal intubation, before pneumoperitoneum, during the first 30 minutes (at 10, 20 and 30 min) of pneumoperitoneum, after release of pneumoperitoneum and 10 min after extubation in the PACU
mean values of heart rate (HR) | 4 hours
  mean values of HR at pre-operative baseline, before induction of anesthesia, 5min after endotracheal intubation, before pneumoperitoneum, during the first 30 minutes (at 10, 20 and 30 min) of pneumoperitoneum, after release of pneumoperitoneum and 10 min after extubation in the PACU
total dose of pethidine given to the patient | 12 hours
  total dose of pethidine given in milligrams will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Ain-Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No